CLINICAL TRIAL: NCT01947465
Title: A Prospective Cohort Study in 6 Swiss Rheumatology Centres and 4 Travel Clinics on the Immunogenicity and Safety of Tetanus and Hepatitis A Vaccine in Patients With Rheumatoid Arthritis, Axial Spondyloarthritis and Vasculitis and Healthy Controls
Brief Title: Immunogenicity and Safety of Vaccinations in Immunocompromised Persons
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: University of Basel (Other); Swiss Tropical & Public Health Institute (Other); University of Bern (Other); University Hospital, Geneva (Other); Cantonal Hospital of St. Gallen (Other); Cantonal Hospital of Aarau, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: CS_2013_01
Record Dates: First submitted 2013-08-22; First posted 2013-09-20 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Arthritis, Rheumatoid; Spondylarthritis; Vasculitis
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylarthritis; Vasculitis | interventions — Hepatitis A Vaccines; Tetanus Toxoid; epaxal berna; Boostrix

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sera from participants will be kept in a biobank for further measurements of antibody responses after vaccination.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Healthy controls: If a vaccination is indicated according to the recommendations by the Swiss Federal Office of Public Health: 319 healthy controls will be enrolled and will receive hepatitis A and/or tetanus vaccination
  Interventions: Biological: Hepatitis A vaccine and tetanus vaccine
- Patients with rheumatoid arthritis: If a vaccination is indicated according to the recommendations by the Swiss Federal Office of Public Health: 142 patients with rheumatoid arthritis will be enrolled and will receive hepatitis A and/or tetanus vaccination.
  Interventions: Biological: Hepatitis A vaccine and tetanus vaccine
- Patients with axial spondylarthritis: If a vaccination is indicated according to the recommendations by the Swiss Federal Office of Public Health: 142 patients with axial spondylarthritis will be enrolled and will receive hepatitis A and/or tetanus vaccination.
  Interventions: Biological: Hepatitis A vaccine and tetanus vaccine
- Patients with vasculitis: If a vaccination is indicated according to the recommendations by the Swiss Federal Office of Public Health: 142 patients with vasculitis will be enrolled and will receive hepatitis A and/or tetanus vaccination.
  Interventions: Biological: Hepatitis A vaccine and tetanus vaccine

INTERVENTIONS:
Biological: Hepatitis A vaccine and tetanus vaccine — Hepatitis A and/or tetanus vaccination will be given to participants in all group on day 0. All monovalent active hepatitis A vaccinations and all vaccines containing tetanus toxoid available in Switzerland may be used in the study
  Other Names: Havrix 1440; Epaxal; Td-Pur; Boostrix; BoostrixPolio; Revaxis

SUMMARY:
Backgound and relevance of the project:

Patients with autoimmune inflammatory rheumatic diseases (AIIRD) are at increased risk of contracting infections. The increased risk can be attributed to the immunological disorder itself, as well as to the immunosuppressive treatment. Vaccination against many infections is recommended in this patient group. However, the immunogenicity of vaccines may be reduced and may also be influenced by the administered treatment. Potential reactivation of the underlying disease triggered by vaccination is another important concern.

From the patients' and public health perspectives, an important task of physicians is giving advice on vaccines. Completing this task is often difficult, because data on the immunogenicity and safety of vaccines in these patient groups are scarce, especially with regard to treatment with new immunosuppressive medications, such as biological agents. Lastly and importantly, due to new therapeutic options, health among AIIRD patients has considerably improved and an increasing number of patients undertake overseas travel activities requiring additional vaccinations. In this context, reliable advice with regard to vaccinations is almost impossible, because for most travel vaccinations the immunogenicity and safety profile is unknown.

Research addressing the immunogenicity and safety of vaccines in different autoimmune inflammatory diseases treated with different immunosuppressive medications is urgently needed to allow giving evidence based vaccine advice.

In this observational study the immunogenicity and safety of tetanus booster and hepatitis A vaccinations will be assessed in AIIRD patients. The immune response will be evaluated as a function of the underlying disease and the possible influence of commonly used immunosuppressive drugs on the immune response will be studied.

Rationale for studying tetanus booster and hepatitis A vaccine Tetanus vaccination is one of the most frequently recommended vaccinations, and the effect of a booster vaccination can be addressed. Hepatitis A vaccine is the most widely used travel vaccine. Despite their importance, only very limited data are available for tetanus and hepatitis A vaccine in this patient group. By focusing on these vaccines the study will lead the way to the evaluation of further vaccines.

The purpose of this study is to determine whether tetanus and hepatitis A vaccinations are as immunogenic and safe in AIIRD patients as in healthy controls.

DETAILED DESCRIPTION:
The study will be placed in 6 rheumatology clinics in Switzerland and in 4 travel medicine clinics. Consecutive subjects with rheumatoid arthritis, spondylarthritis (ankylosing spondylitis), vasculitis (ANCA associated vasculitis and Behçet's disease) and healthy controls will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Indication for hepatitis A and/or tetanus vaccination according to Swiss Federal Office of Public Health recommendations
* Male and female rheumatic patients with rheumatoid arthritis or axial spondyloarthritis (ankylosing spondylitis, axial psoriatic arthritis, axial undifferentiated spondyloarthritis, enteropahtic arthritis) or peripheral psoriatic arthritis or vasculitis (Behçet's disease or ANCA-associated vasculitis) or male and female healthy participants ≥ 18 years
* Signed Informed Consent after being informed

Exclusion Criteria:

* Known hypersensitivity to a vaccine ingredient
* Estimated patient survival below 1 year
* Active malignant or active infectious disease
* Drug/alcohol abuse
* Insufficient understanding of local language

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The cohort will be selected from patients with rheumatic diseases under treatment at 6 rheumatology outpatient clinics in Switzerland (University of Basel, University of Bern, University of Geneva, University of Zurich, Cantonal Hospital Aarau, Cantonal Hospital St. Gallen)
Sampling Method: Probability Sample
Enrollment: 645 (Actual)
Dates: Start 2013-10; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Immunogenicity of hepatitis A and tetanus vaccination in patients with rheumatoid arthritis, axial spondyloarthritis and vasculitis and in healthy controls | Change from Baseline in geometric mean antibody titre and seroprotection at 4 weeks and at 12 weeks
  comparison of the geometric mean antibody titre and percentage of seroprotected individuals after tetanus and hepatitis A vaccination between each disease group and healthy controls

SECONDARY OUTCOMES:
Safety of tetanus and hepatitis A vaccines in patients with rheumatoid arthritis, axial spondyloarthritis and vasculitis and in healthy controls | Activation of rheumatic disease will be assessed for 1 week after vaccine administration and at 4 and 12 weeks compared to baseline
  Number of patients with any worsening or reactivation of the rheumatic disease after vaccine administration
  Number of participants with adverse vaccine reactions (local and systemic reactions) in patients with rheumatoid arthritis, axial spondyloarthritis and vasculitis and in healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Hatz, Professor, Principal Investigator — University of Zurich
Locations (10):
- Switzerland (10):
  - University Hospital of Basel, Rheumatology Division, Basel, Basel Town
  - Swiss Tropical and Public Health Institute, Basel, Basel Town
  - Cantonal Hospital Aarau, Division of Rheumatology, Aarau, Canton of Aargau
  - University of Bern, Inselspital, Division of Infectious Diseases and Travel Medicine, Bern, Canton of Bern
  - University of Bern, Inselspital, Division of Rheumatology, Bern, Canton of Bern
  - University of Geneva, University Hospitals, Division of Rheumatology, Geneva, Canton of Geneva
  - University of Geneva, University Hospitals, Service de Médecine Tropicale et Humanitaire, Geneva, Canton of Geneva
  - Cantonal Hospital St. Gallen, Division of Rheumatology, Sankt Gallen, Canton of St. Gallen
  - University of Zurich, Epidemiology, Biostatistics and Prevention Institute, Divison of Infectious Diseases, Zurich, Canton of Zurich
  - University of Zurich, University Hopsital, Divison of Rheumatology, Zurich, Canton of Zurich

REFERENCES:
- [Background] van Assen S, Elkayam O, Agmon-Levin N, Cervera R, Doran MF, Dougados M, Emery P, Geborek P, Ioannidis JP, Jayne DR, Kallenberg CG, Muller-Ladner U, Shoenfeld Y, Stojanovich L, Valesini G, Wulffraat NM, Bijl M. Vaccination in adult patients with auto-immune inflammatory rheumatic diseases: a systematic literature review for the European League Against Rheumatism evidence-based recommendations for vaccination in adult patients with auto-immune inflammatory rheumatic diseases. Autoimmun Rev. 2011 Apr;10(6):341-52. doi: 10.1016/j.autrev.2010.12.003. Epub 2010 Dec 20. PMID 21182987
- [Background] Bijl M, Kallenberg CG, van Assen S. Vaccination of the immune-compromised patients with focus on patients with autoimmune-inflammatory diseases. Neth J Med. 2011 Jan;69(1):5-13. PMID 21325695
- [Background] Doran MF, Crowson CS, Pond GR, O'Fallon WM, Gabriel SE. Frequency of infection in patients with rheumatoid arthritis compared with controls: a population-based study. Arthritis Rheum. 2002 Sep;46(9):2287-93. doi: 10.1002/art.10524. PMID 12355475
- [Background] Bernatsky S, Hudson M, Suissa S. Anti-rheumatic drug use and risk of serious infections in rheumatoid arthritis. Rheumatology (Oxford). 2007 Jul;46(7):1157-60. doi: 10.1093/rheumatology/kem076. Epub 2007 May 3. PMID 17478469
- [Background] Kotton CN. Vaccination and immunization against travel-related diseases in immunocompromised hosts. Expert Rev Vaccines. 2008 Jul;7(5):663-72. doi: 10.1586/14760584.7.5.663. PMID 18564020
- [Background] Rahier JF, Moutschen M, Van Gompel A, Van Ranst M, Louis E, Segaert S, Masson P, De Keyser F. Vaccinations in patients with immune-mediated inflammatory diseases. Rheumatology (Oxford). 2010 Oct;49(10):1815-27. doi: 10.1093/rheumatology/keq183. Epub 2010 Jun 29. PMID 20591834
- [Background] Steffen R, Kane MA, Shapiro CN, Billo N, Schoellhorn KJ, van Damme P. Epidemiology and prevention of hepatitis A in travelers. JAMA. 1994 Sep 21;272(11):885-9. PMID 8078167
- [Background] Agarwal N, Ollington K, Kaneshiro M, Frenck R, Melmed GY. Are immunosuppressive medications associated with decreased responses to routine immunizations? A systematic review. Vaccine. 2012 Feb 14;30(8):1413-24. doi: 10.1016/j.vaccine.2011.11.109. Epub 2011 Dec 21. PMID 22197580
- [Derived] Buhler S, Jaeger VK, Adler S, Bannert B, Brummerhoff C, Ciurea A, Distler O, Franz J, Gabay C, Hagenbuch N, Herzog C, Hasler P, Kling K, Kyburz D, Muller R, Nissen MJ, Siegrist CA, Villiger PM, Walker UA, Hatz C. Safety and immunogenicity of tetanus/diphtheria vaccination in patients with rheumatic diseases-a prospective multi-centre cohort study. Rheumatology (Oxford). 2019 Sep 1;58(9):1585-1596. doi: 10.1093/rheumatology/kez045. PMID 30877773
- See also: Vaccination recommendations in immunocompromised travelers by the Centers for Disease Control and Prevention — http://wwwnc.cdc.gov/travel/yellowbook/2014/chapter-8-advising-travelers-with-specific-needs/immunocompromised-travelers
- See also: Vaccination recommendations in immunocompromised persons, Belgium — http://www.health.belgium.be/internet2Prd/groups/public/@public/@shc/documents/ie2divers/19080078_en.pdf
- See also: Vaccination recommendation for patients with rheumatic disease, Swiss society of rheumatology — http://www.rheuma-net.ch/download/Content_attachments/FileBaseDoc/Impfempfehlungen-D.pdf